CLINICAL TRIAL: NCT05881876
Title: Determining the Reliability and Validity of a New Method for Measuring Upper Extremity Joint Range of Motion in Burn Patients Using a Tracking System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, So Young Joo, Hangang Sacred Heart Hospital, Hangang Sacred Heart Hospital
Other Study IDs: HangangSHH-14
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Contracture Joint

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- burn groups: Inclusion criteria were as follows: male or female patients between 18 and 75 years of age, partial or full-thickness burns that healed spontaneously or required skin grafting, and limited joint ROM in the upper extremities caused by burns.

SUMMARY:
In burn patients, joint contracture is a common complication caused by hypertrophic scars, necessitating accurate evaluation and diagnosis of the degree of disability and functional deterioration. A standard goniometer based on the American Medical Association (AMA) guidelines for measuring joint range of motion (ROM) is the gold standard for evaluating musculoskeletal diseases. However, the handheld goniometer is highly dependent on the skill and experience of the measurer. Recently, a marker-based system for accurate ROM measurement has been demonstrated in clinical evaluation. This study investigated the reliability and validity of the marker-based system for evaluation of joint ROM in burn patients.

Inclusion criteria were as follows: male or female patients between 18 and 75 years of age, partial or full-thickness burns that healed spontaneously or required skin grafting, and limited joint ROM in the upper extremities caused by burns. Exclusion criteria were limited joint ROM due to severe osteoarthritis or rheumatoid arthritis, congenital defects, structural disease, amputation, central or peripheral nervous system injuries, difficulty in voluntary decision-making due to cognitive impairment, or a history of orthopaedic surgery due to fracture.

The experimentals tried to compare the validity and reliability of a marker-based system and AMA methods for the burn patient with joint contracture of upper extremities.

DETAILED DESCRIPTION:
In burn patients, joint contracture is a common complication caused by hypertrophic scars, necessitating accurate evaluation and diagnosis of the degree of disability and functional deterioration. A standard goniometer based on the American Medical Association (AMA) guidelines for measuring joint range of motion (ROM) is the gold standard for evaluating musculoskeletal diseases. However, the handheld goniometer is highly dependent on the skill and experience of the measurer. Recently, a marker-based system for accurate ROM measurement has been demonstrated in clinical evaluation. This study investigated the reliability and validity of the marker-based system for evaluation of joint ROM in burn patients.

After three familiarisation trials for ROM measurement, the evaluation procedure was initiated on the participant's dominant side. A standard goniometer was used to measure ROM and increments were marked. The measurement position was the same as that used in the standard Korean range of motion protocol (KRSP). One examiner measured aROM for flexion, extension, abduction, adduction, external rotation, and internal rotation at a neutral position using a stainless-steel goniometer (JAMAR Co., Pakistan). The aROM was measured under the instruction that the subjects should move their arms as far as possible.

For ROM evaluation in upper extremities, 22 reflective markers were attached to the patient's body before measurement and markers were tracked using eight infrared cameras. Prior to the test, a static calibration test was performed in a neutral position. A skeleton model was obtained directly from the Motive2.1 (the unified software platform of OptiTrack®) for the data gathered by the OptiTrack® system (NaturalPoint, Inc., Corvallis, OR, USA). The ROM of the shoulder, elbow, and wrist was measured sequentially using a dynamic view. The marker trajectories allowed estimation of the joint centres and definition. The joint centres were calculated from optical motion capture data, according to the definitions of Visual3D (C-Motion, Inc., Germantown, MD, USA), a widely used software tool for 3D biomechanical research.

After evaluating the ROM of the upper extremity joint using a goniometer and optical motion capture system (session 1), re-measurement was performed 2 days later (session 2). Markers were positioned by the same observer in both sessions for all the participants.

All statistical analyses were performed using SPSS version 23 (IBM Corp., Armonk, NY, USA). The mean ROM and standard deviation were calculated. An independent t-test was used to compare inter-method differences. For intra-rater reliability, two tests were compared for each measurement. Relative reliability was assessed using the intraclass correlation coefficient (ICC) and ICC interpretation was based on the Fleiss guidelines. Statistical significance was set as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* ages between 18 and 75 years of age
* partial or full-thickness burns that healed spontaneously or required skin grafting
* limited joint ROM in the upper extremities caused by burns.

Exclusion Criteria:

* limited joint ROM due to severe osteoarthritis or rheumatoid arthritis
* congenital defects, structural disease, amputation
* central or peripheral nervous system injuries
* difficulty in voluntary decision-making due to cognitive impairment
* a history of orthopaedic surgery due to fracture.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: who had developed joint contractures in the shoulder, elbow or wrist due to hypertrophic scars after thermal injury were enrolled in this study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
range of motion of joint | 2 days
  For ROM evaluation in upper extremities, 22 reflective markers were attached to the patient's body before measurement and markers were tracked using eight infrared cameras. Prior to the test, a static calibration test was performed in a neutral position. A skeleton model was obtained directly from the Motive2.1 (the unified software platform of OptiTrack®) for the data gathered by the OptiTrack® system (NaturalPoint, Inc., Corvallis, OR, USA).The ROM of the shoulder, elbow, and wrist was measured sequentially using a dynamic view. The marker trajectories allowed estimation of the joint centres and definition (Figure 1). The joint centres were calculated from optical motion capture data, according to the definitions of Visual3D (C-Motion, Inc., Germantown, MD, USA), a widely used software tool for 3D biomechanical research .

SECONDARY OUTCOMES:
AMA evaluation | 2 days
  A standard goniometer was used to measure ROM and increments were marked. The measurement position was the same as that used in the standard Korean range of motion protocol (KRSP). One examiner measured aROM for flexion, extension, abduction, adduction, external rotation, and internal rotation at a neutral position using a stainless-steel goniometer (JAMAR Co., Pakistan). The aROM was measured under the instruction that the subjects should move their arms as far as possible.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schouten HJ, Nieuwenhuis MK, van Baar ME, van der Schans CP, Niemeijer AS, van Zuijlen PPM. The degree of joint range of motion limitations after burn injuries during recovery. Burns. 2022 Mar;48(2):309-318. doi: 10.1016/j.burns.2021.01.003. Epub 2021 Jan 22. PMID 34955294
- [Background] Ahn SY, Ko H, Yoon JO, Cho SU, Park JH, Cho KH. Determining the Reliability of a New Method for Measuring Joint Range of Motion Through a Randomized Controlled Trial. Ann Rehabil Med. 2019 Dec;43(6):707-719. doi: 10.5535/arm.2019.43.6.707. Epub 2019 Dec 31. PMID 31918533